CLINICAL TRIAL: NCT05264701
Title: Investigation of the Effects of Artificial Intelligence-supported and Technology-based Cardiac Rehabilitation Programs on Participation and Exercise Capacity in Coronary Artery Patients
Brief Title: Investigation of the Effects of the Technology-based Cardiac Rehabilitation Program in Coronary Artery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Saklica, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-20105
Record Dates: First submitted 2022-02-19; First posted 2022-03-03 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease; Physical Inactivity
Keywords: Cardiac Rehabilitation; Exercise Training
MeSH Terms: conditions — Coronary Artery Disease; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapist Supervised Exercise Training Group (Experimental): Physiotherapist supervised exercise training in patients with coronary artery disease
  Interventions: Other: Physiotherapist supervised exercise training
- Exercise Training Tracking from Phone-app Group (Experimental): Exercise training tracking from phone app in patients with coronary artery disease
  Interventions: Other: Exercise training via phone app
- Control Group (Experimental): General physical activity recommendations for home
  Interventions: Other: Physical activity recommendations

INTERVENTIONS:
Other: Physiotherapist supervised exercise training — Exercise training for 12 weeks will be given by video talk accompanied by a physiotherapist.
  Arms: Physiotherapist Supervised Exercise Training Group
Other: Exercise training via phone app — Exercise training for 12 weeks will be given over the developed phone application.
  Arms: Exercise Training Tracking from Phone-app Group
Other: Physical activity recommendations — The program will be consist of 12 weeks of physical activity recommendations.
  Arms: Control Group

SUMMARY:
This study was planned to investigate the effectiveness of technology-based and traditional cardiac rehabilitation programs in individuals with coronary artery disease.

DETAILED DESCRIPTION:
Cardiovascular diseases constitute one of the most critical health problems of today's society due to the loss of workforce, morbidity, mortality, and high hospital expenses.

This study was planned to investigate the effectiveness of technology-based and traditional cardiac rehabilitation programs in individuals with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease
* Access to the online program
* Volunteering to participate in the research
* Having an iOS or Android operating system compatible phone

Exclusion Criteria:

* Having a musculoskeletal problem
* Having uncontrolled hypertension
* Having chronic heart failure (NYHA III-IV)
* A history of acute coronary syndrome or surgical revascularization less than 12 months ago
* More than 50% occlusion on the main coronary artery
* Having arrhythmia

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Baseline, after 12 weeks, after 24 weeks
  Exercise capacity will be evaluated using the incremental shuttle walk test.
Participation | after 12 weeks
  Participation will be evaluated using the number of sessions attended.

SECONDARY OUTCOMES:
Maximal Effort Capacity | Baseline
  Maximal effort capacity will be evaluated using a cardiovascular stress test.
Peripheral muscle strength | Baseline, after 12 weeks, after 24 weeks
  Peripheral muscle strength will be evaluated using the dynamometer.
Endothelial function | Baseline, after 12 weeks, after 24 weeks
  The endothelial function will be evaluated using echocardiography. After a resting baseline, Brachial artery diameter will be recorded, the cuff used in blood pressure measurement will be inflated 25-50 mmHg above the systolic blood pressure value and maintain that pressure for 5 min. The brachial artery diameter will be measured again after the cuff is deflated.
Healthy Living Habit Evaluation | Baseline, after 12 weeks, after 24 weeks
  Healthy living habit evaluation will be evaluated using the Healthy Lifestyle Behaviors Scale-II.
Health-Related Quality of Life | Baseline, after 12 weeks, after 24 weeks
  Health-Related Quality of Life will be evaluated using the Myocardial Infarction Dimensional Assessment Scale (MIDAS).
QoL | Baseline, after 12 weeks, after 24 weeks
  Quality of life will be evaluated using the SF-36 Short Form.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Hikmet Yorgun, PhD, Study Director — Hacettepe University; Ahmet Hakan Ates, PhD, Study Chair — Hacettepe University; Deniz Yuce, PhD, Study Chair — Hacettepe University; Dilara Saklica, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)